CLINICAL TRIAL: NCT04441801
Title: Optimal Duration of Stretching of the Hamstring Muscle Group : A Randomized Controlled Trial
Brief Title: Optimal Duration of Stretching of the Hamstring Muscle Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Principal Investigator, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USharjah
Record Dates: First submitted 2020-06-12; First posted 2020-06-22 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Physical and Rehabilitation Medicine
Keywords: Stretching; Randomized controlled trial; Hamstring
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: A prospective, parallel-group, randomized clinical trial participants will be randomly assigned to the control group or one of the 3 intervention groups .The three experimental groups was stretched for 15, 30, and 60 seconds, respectively the control group did not stretch
Who Masked: Outcomes Assessor
Masking Description: The assessor, who took the measurements for both the intervention and control groups, was blinded to the subject's group, while the treating therapist was not blinded to the treatment intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 15 seconds (Experimental): Stretching of the hamstring muscles will be performed by the primary researcher. A straight-leg-raising technique will be used for this stretch because we believe that it is commonly used in the clinical setting for elderly people. All subjects were supine lying as flat as possible, each subject's knee will be maintained in extension with the ankle at 90 degrees without medial (internal) or lateral (external) rotation of the lower extremity, and the extremity was raised until the subject reported discomfort. The subject was asked to relax the lower extremity in an effort to prevent contracting muscles from affecting the stretch and to allow for a slow stretch. stretching will continue for 15 seconds .The patient relaxed for approximately 20s and the procedure was repeated three times.
  Interventions: Other: stretching exercise
- 30 seconds (Experimental): the same stretching technique will continue for 30 seconds .The patient relaxed for approximately 20s and the procedure was repeated three times.
  Interventions: Other: stretching exercise
- 60 seconds (Experimental): the same stretching technique will continue for 60 seconds .The patient relaxed for approximately 20s and the procedure was repeated three times.
  Interventions: Other: stretching exercise
- control (Sham Comparator): The control group followed the same procedures except that no stretching force was applied at the end.
  Interventions: Other: stretching exercise

INTERVENTIONS:
Other: stretching exercise — Static stretching consists of stretching a muscle (or group of muscles) to its farthest point and then maintaining or holding that position

SUMMARY:
OBJECTIVE: To explore the effect of variable stretching intervals on neural function and ROM.

DESIGN: Randomized controlled trial Participants: In this trial, 168 participants diagnosed with tight hamstring muscles (defined as the inability to extend the knee to less than 20° of knee flexion) were randomly assigned to the control group or one of the 3 intervention groups Interventions: The three experimental groups was stretched for 15, 30, and 60 seconds, respectively the control group did not stretch Main Outcome Measures: The neurophysiological outcome measures included peak to peak somatosensory evoked potential for dermatomes L3,L4,L5, and S1. Secondary outcome measures included knee ROM. All outcome measures were assessed immediately after the treatment session and 24 hours after the treatment session.

DETAILED DESCRIPTION:
A prospective, blinded, parallel-group, randomized clinical trial will be conducted in the research laboratory of our university. The patients will participate in the study after signing an informed consent form prior to data collection.

Inclusion Criteria Subjects who demonstrate "tight" hamstring muscles, defined as inability to extend the knee to less than 20 degrees of knee flexion with the femur held at 90 degrees of hip flexion while the person was positioned supine. Subjects will also be screened to rule out knee joint flexion contractures by checking knee extension ROM, while they were lying in a prone position Exclusion Criteria Using of medical aids, and suffering from any neurological or cognitive impairment, limiting cardio-respiratory conditions, or had undergone recent surgery (within the past 12 months). Having any hip or knee replacements or any history of pathology in the low back, hips, or knees for the 3 months prior to the study

Participants will be divided into four groups according to the stretching duration time (15, 30, and 60s, and the fourth group, which served as a control, did not stretch). The patients will randomly assigned to one of the four groups as follows. The randomization process will be based on permuted blocks of variable sizes. Each random permuted block, created randomly by a number generator, will be transferred to a sequence of consecutively numbered, opaque, sealed envelopes that will be kept in a locked drawer until needed. Once a subject was formally included in the trial, the next envelope in the sequence was opened by the researcher in the presence of the subject who would be assigned to a group according to the number found in the envelope.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with "tight" hamstring muscles, defined as inability to extend the knee to less than 20 degrees of knee flexion with the femur held at 90 degrees of hip flexion while the person was positioned supine.

Exclusion Criteria:

* Using of medical aids.
* suffering from any neurological or cognitive impairment, limiting cardio-respiratory conditions,
* had undergone recent surgery (within the past 12 months).
* Having any hip or knee replacements or any history of pathology in the low back, hips, or knees for the 3 months prior to the study

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Change in dermatomal somatosensory evoked potentials immediately after treatment | pre-treatment , immediately after treatment and at 24 hours after the treatment .
  In all dermatomes, 2 complete recording runs will be undertaken during each session with averages of 250 to 1200 cortical responses from scalp surface recording electrodes (C3'-C4' in a 10-20 electrode configuration) of the contralateral scalp to the stimulated dermatomes being stimulated. The impedance of ground and scalp electrodes will be maintained at < 5 k Cutaneous areas of L3,L4,L5, S1 sensory roots will be stimulated in lower limb with the electrical impulses of 0.2 ms duration, frequency of 3.3 Hz and intensity 3 times higher than the sensory threshold will be determined individually for each subject.

SECONDARY OUTCOMES:
change in range of motion | pre-treatment , immediately after treatment and at 24 hours after the treatment .
  Each subject will then be measured for knee extension ROM . Measurement of knee extension ROM was made with the subject lying supine with the opposite lower extremity extended and the lower extremity being measured positioned at 90 degrees of hip flexion. The greater trochanter and the lateral epicondyle of the femur and lateral malleolus will be palpated and served as landmarks during measurement, The measurement recorded will be the angle between the leg position and full knee extension (considered to be 0°). Because knee joint contractures will be ruled out, the measurement of knee extension ROM was considered to be an indirect measure of hamstring muscle flexibility, with hamstring muscle tightness being the purported cause of a lack of knee extension ROM.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Moustafa, professor, Principal Investigator — University of Sharjah
Locations (1):
- Ibrahim Moustafa, Sharjah city, United Arab Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data (IPD) available to other researchers.